CLINICAL TRIAL: NCT03820882
Title: Catfish Flow Restoration Device for Thrombectomy Revascularisation of Large Vessel Occlusions in Acute Ischemic Stroke: a Randomised, Parallel-group, Non-inferiority Trial
Brief Title: Stent Retriever for Thrombectomy Revascularisation of Large Vessel Occlusions in Acute Ischemic Stroke(Catfish)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Zhongrong Miao, Director, Head of Neurointerventional, Principal Investigator, Clinical Professor, Ministry of Science and Technology of the People´s Republic of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JSSKBMCT001
Record Dates: First submitted 2019-01-14; First posted 2019-01-29 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: prospective, randomized, open-label, parallel assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stent retriever(Catfish) (Experimental): Mechanical thrombectomy with Catfish flow restoration device
  Interventions: Device: Catfish
- stent retriever(Solitaire FR) (Active Comparator): Mechanical thrombectomy with Solitaire FR flow restoration device
  Interventions: Device: Solitaire FR

INTERVENTIONS:
Device: Catfish — Patients will be treated for mechanical recanalization with Catfish within 8 hours after stroke onset plus standard medical management.
  Arms: stent retriever(Catfish)
Device: Solitaire FR — Patients will be treated for mechanical recanalization with Solitaire FR within 8 hours after stroke onset plus standard medical management.
  Arms: stent retriever(Solitaire FR)

SUMMARY:
The study is a randomized, prospective, parallel-group, multicenter, open-label, non-inferiority trial. Patients are randomized 1 : 1 to either stent retriever(Catfish) or Solitaire for endovascular therapy for acute ischemic stroke. The study aims to evaluate the benefit and safety of stent retriever(Catfish) for acute ischemic stroke therapy, as compared to Solitaire FR.

DETAILED DESCRIPTION:
The main objective is to determine whether stent retriever(Catfish) will have non-inferior successful recanalization rate compared to Solitaire in patients with acute ischemic stroke caused by large vessel occlusion.

The secondary objectives is to verify whether there is significant differences in time from artery puncture to successful recanalization (mTICI 2b or greater), NIHSS score at 24 hours and at 7 days or discharge if earlier, good clinical outcomes at 90 days (defined as mRS score ≤2) between stent retriever(Catfish) and Solitaire in patients with acute ischemic stroke caused by large vessel occlusion.

The third objectives is to compare the rate of symptomatic intracranial hemorrhage, serious adverse event(SAE), all cause of mortality with 90 days after operation, between stent retriever (Catfish) and Solitaire in patients with acute ischemic stroke due to large vessel occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ages≤80;
2. mRS score must lower than 2 Pre-AIS(acute ischemic stroke).
3. Baseline NIHSS score obtained prior to randomization must be between 8 and 25;
4. Symptoms and signs in accordance with Large vessel occlusion, confirmed by CTA(CT angiogram)/MRA(magnetic resonance angiography )/DSA;
5. Patient treatable within 8 hours of symptom onset (symptoms onset is defined as point in time the patient was last seen well (at baseline)) can accept the complete femoral artery puncture;
6. Baseline Alberta stroke program early CT score (ASPECTS) or posterior circulation Alberta stroke program early CT score (pc-ASPECTS)≥ 6 on Computed tomography (CT) or magnetic resonance imaging(MRI).
7. The patient or relative give written informed consent.

Exclusion Criteria:

1. History of stroke in past 3 months.
2. Presumed septic embolus, or suspicion of bacterial endocarditis.
3. Evidence of tortuosity of cervical vessels precluding device delivery/deployment;
4. Hypertension (Systolic blood pressure(SBP)>185 mmHg or diastolic blood pressure(DBP)>110 mm Hg) after using drug;
5. Platelet count<30,000/μL and use of Novel Anticoagulant with International Normalized Ratio(INR)>3.0;
6. Random blood glucose of<2.7mmol/L or>22.2mmol/L;
7. Patients with heart or lung or liver or renal failure or other sever disease (intracranial tumors, cerebral arteriovenous malformation (AVM), systemic infection, active disseminated intravascular coagulation, history of sever psychosis);
8. Patients with Dementia or psychiatric disease that would confound the neurological or functional evaluations.
9. Anticipated life expectancy of less than 6 months;
10. Known serious sensitivity to contrast medium and nitinol metal;
11. Females who are pregnant or breastfeeding;
12. Current participation in any other clinical trial;
13. The patient or the patient's legally authorized representative hasn't signed and dated an informed consent form;
14. Rapidly improving neurologic examination.
15. Excessive vascular access tortuosity that will likely result in unstable access platform.
16. Seizures at stroke onset which would preclude obtaining a baseline NIHSS.
17. Suspected intracranial dissection or cerebral vasculitis.
18. Evidence of tandem cervical occlusion, or stenosis requiring treatment.
19. Major surgery or significant trauma in the past 30 days or plan to have surgery in next 3 months after enrolled.
20. CT or MRI evidence of mass effect or intra-cranial tumour (except small meningioma)
21. Any type of cerebral hemorrhage (only microbleeds are allowed) on neuroimaging
22. The subject is not appropriate for mechanical thrombectomy intervention in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Instant recanalization rate (mTICI 2b-3) of target vessel after the procedure | immediate
  Successful recanalization is defined as modified Thrombolysis In Cerebral Ischemia scale 2b or 3. And it is evaluated by DSA(digital subtraction angiography ) intraoperative immediately in both treatment groups

SECONDARY OUTCOMES:
Time to achieve recanalization | intraprocedure immediate
  The period from femoral artery puncture to successful recanalization
NIHSS score at 24±2 hours | 24±2 hours
  National Institutes of Health Stroke Scale( NIHSS),the NIHSS is a stroke severity score that is composed of 11 items; range from 0 to 42, higher values indicate more severe deficits
NIHSS score at 7±1 days or discharge | 7±1 days
  National Institutes of Health Stroke Scale( NIHSS),the NIHSS is a stroke severity score that is composed of 11 items; range from 0 to 42, higher values indicate more severe deficits
proportion of patients who got a mRS 0-2 at 90±14 days | 90±14 days
  The proportion of patients who got a mRS 0-2 in patients who receive stent retriever treatment.the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death)
symptomatic intracranial hemorrhage after procedure | 24±2 hours
  sICH was defined as any type of ICH on neuroimaging after the treatment within 24±2 hours after procedure with increasing of ≥4 points on NIHSS, National Institutes of Health Stroke Scale( NIHSS),the NIHSS is a stroke severity score that is composed of 11 items; range from 0 to 42, higher values indicate more severe deficits
serious adverse event(SAE) within 90±14 days after procedure | 90±14 days
all cause of mortality within 90±14 days after procedure | 90±14 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Luo G, Yan X, Xiao G, Wei L, Nai Bi Jiang YLK, Ma R, Chen W, Fang C, Zhou Z, Wan J, Peng Y, Zhang G, Zhao J, Li L, Yuan H, Wu J, Li B, Zhang F, Cheng Y, Gao F, Miao Z. Comparing a novel Catfish flow restoration device and the Solitaire stent retriever for thrombectomy revascularisation in emergent largevessel occlusion stroke: a prospective randomised controlled study. Stroke Vasc Neurol. 2023 Dec 29;8(6):435-443. doi: 10.1136/svn-2022-002036. PMID 37045544